CLINICAL TRIAL: NCT03008135
Title: Reliability and Validity of the Elderly Mobility Scale for Frailty People Living at Home, French Version
Brief Title: Reliability and Validity of the Elderly Mobility Scale, French Version
Status: Completed | Type: Observational
Sponsor: Pole Santé Plouasne Saint Pern Becherel (Other)
Responsible Party: Sponsor
Other Study IDs: PSPB-01-2016
Record Dates: First submitted 2016-12-16; First posted 2017-01-02 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Locomotor Activity; Functionally-Impaired Elderly; Frail Elderly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Elderly Mobility Scale — The Elderly Mobility Scale was devised to assess the mobility of fragile elderly people, and contains seven items considered as essential for performing the basic activities of the daily routine: Lying down to sitting, sitting to lying down, sitting to standing, standing, Gait/ work on body posture, timed walk (6 meters) and work on Functional Reach/movements?
Other: Frailty scale — 6 questions are asked to the person about his or her living conditions to determine the level of frailty. The scale is produced by the board "High Health Authority"

SUMMARY:
This study evaluates the reliability of the French version of the "elderly mobility scale" and its correlation with the "frailty elderly scale "

DETAILED DESCRIPTION:
The research question:

How to effectively measure the physical independence of the elderly at home and how, from this measure, the investigators can determine the fragility threshold of the elderly.

The elderly mobility scale measures the critical points of the patient's physical autonomy. This scale was developed in Great Britain. The purpose of this study is to establish the reliability of this French version scale and to study the correlation with the elderly scale fragility.

People are recruited by a Medical consultant. After consent, their frailty is measured and a prescription is done to see a Physical therapist. The physical therapist will evaluate the physical points measured/ mentioned in the Elderly Mobility Scale, twice in a week, with two different assessors.

ELIGIBILITY:
Inclusion Criteria:

* living at home, more than 70 years old

Exclusion Criteria:

* current recovery for orthopaedic problems
* Cognition impairment
* all acute problems with an impairment of mobility

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: People living in their home, more than 70 years old, alone or not.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2017-10-26 (Actual); Study Completion 2017-10-26 (Actual)

PRIMARY OUTCOMES:
inter-rater Reliability | Time Frame: Up to One week
  intraclass correlation coefficient with data : Elderly Mobility Scale score between rater one and rater two

SECONDARY OUTCOMES:
Concurrent Validity | Time Frame: Up to One week
  correlation coefficient between Elderly Mobility Scale and Frailty scale
sensibility and specificity | Time Frame: Up to One week
  sensibility and specificity of Elderly Mobility Scale regarding Frailty
Receiver Operating Curve and cut-off score | Time Frame: Up to One week
  Determination of a cut-off score for Elderly Mobility Scale as a screening tool to detect the frailty by use of Receiver Operating Characteristics curve

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Cabinet medical, Bécherel
  - Cabinet medical, Plouasne
  - Cabinet de kinésithérapie, Saint-Pern

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Crocker T, Forster A, Young J, Brown L, Ozer S, Smith J, Green J, Hardy J, Burns E, Glidewell E, Greenwood DC. Physical rehabilitation for older people in long-term care. Cochrane Database Syst Rev. 2013 Feb 28;2013(2):CD004294. doi: 10.1002/14651858.CD004294.pub3. PMID 23450551
- [Background] Lihavainen K, Sipila S, Rantanen T, Kauppinen M, Sulkava R, Hartikainen S. Effects of comprehensive geriatric assessment and targeted intervention on mobility in persons aged 75 years and over: a randomized controlled trial. Clin Rehabil. 2012 Apr;26(4):314-26. doi: 10.1177/0269215511423269. Epub 2011 Oct 17. PMID 22007041
- [Background] Daniels R, Metzelthin S, van Rossum E, de Witte L, van den Heuvel W. Interventions to prevent disability in frail community-dwelling older persons: an overview. Eur J Ageing. 2010 Feb 9;7(1):37-55. doi: 10.1007/s10433-010-0141-9. eCollection 2010 Mar. PMID 28798616
- [Background] Clegg A, Barber S, Young J, Forster A, Iliffe S. The Home-Based Older People's Exercise (HOPE) trial: study protocol for a randomised controlled trial. Trials. 2011 Jun 8;12:143. doi: 10.1186/1745-6215-12-143. PMID 21651805
- [Background] Clegg AP, Barber SE, Young JB, Forster A, Iliffe SJ. Do home-based exercise interventions improve outcomes for frail older people? Findings from a systematic review. Rev Clin Gerontol. 2012 Feb;22(1):68-78. doi: 10.1017/S0959259811000165. Epub 2012 Aug 24. PMID 27226701
- [Background] Morley JE, Vellas B, van Kan GA, Anker SD, Bauer JM, Bernabei R, Cesari M, Chumlea WC, Doehner W, Evans J, Fried LP, Guralnik JM, Katz PR, Malmstrom TK, McCarter RJ, Gutierrez Robledo LM, Rockwood K, von Haehling S, Vandewoude MF, Walston J. Frailty consensus: a call to action. J Am Med Dir Assoc. 2013 Jun;14(6):392-7. doi: 10.1016/j.jamda.2013.03.022. PMID 23764209
- [Background] Guralnik JM, Ferrucci L, Simonsick EM, Salive ME, Wallace RB. Lower-extremity function in persons over the age of 70 years as a predictor of subsequent disability. N Engl J Med. 1995 Mar 2;332(9):556-61. doi: 10.1056/NEJM199503023320902. PMID 7838189
- [Background] Shumway-Cook A, Brauer S, Woollacott M. Predicting the probability for falls in community-dwelling older adults using the Timed Up & Go Test. Phys Ther. 2000 Sep;80(9):896-903. PMID 10960937
- [Background] Downs S, Marquez J, Chiarelli P. Normative scores on the Berg Balance Scale decline after age 70 years in healthy community-dwelling people: a systematic review. J Physiother. 2014 Jun;60(2):85-9. doi: 10.1016/j.jphys.2014.01.002. Epub 2014 Jun 13. PMID 24952835
- [Background] C. for R. O. R. Rehabilitation Institute of Chicago, " Rehab Measures : Barthel Index Rehabilitation Measures Database ", 2014. [En ligne]. Disponible sur: http://www.rehabmeasures.org/Lists/RehabMeasures/PrintView.aspx?ID=916.
- [Background] Karpman C, Lebrasseur NK, Depew ZS, Novotny PJ, Benzo RP. Measuring gait speed in the out-patient clinic: methodology and feasibility. Respir Care. 2014 Apr;59(4):531-7. doi: 10.4187/respcare.02688. Epub 2013 Aug 27. PMID 23983271
- [Background] Stineman MG, Shea JA, Jette A, Tassoni CJ, Ottenbacher KJ, Fiedler R, Granger CV. The Functional Independence Measure: tests of scaling assumptions, structure, and reliability across 20 diverse impairment categories. Arch Phys Med Rehabil. 1996 Nov;77(11):1101-8. doi: 10.1016/s0003-9993(96)90130-6. PMID 8931518
- [Background] C. Flahault, C. Généraux, A. Colvez, V. Royer, et S. Berthié-mourgaud, " ETUDE DE LA FIABILITE DE L ' INSTRUMENT AGGIR Reproductibilité ( test / re-test ) entre évaluateurs Dispersion des temps d ' aide requise entre Groupes Iso Ressources Enquête dans cinq départements Travail réalisé par Dans l ' Hérault Dans les Alpes marit ", 2005
- [Background] S. C. B. Ennie, K. A. B. Runer, et A. L. D. Izon, " Measurements of Balance : Comparaison of the Timed "up and Go" Test and Functional Reach Test with the Berg Balance Scale ", J. Phys. Ther. Sci., vol. 15, p. 93-97, 2003.
- [Background] Yu MS, Chan CC, Tsim RK. Usefulness of the Elderly Mobility Scale for classifying residential placements. Clin Rehabil. 2007 Dec;21(12):1114-20. doi: 10.1177/0269215507080789. PMID 18042607
- [Result] Rolland Y, Benetos A, Gentric A, Ankri J, Blanchard F, Bonnefoy M, de Decker L, Ferry M, Gonthier R, Hanon O, Jeandel C, Nourhashemi F, Perret-Guillaume C, Retornaz F, Bouvier H, Ruault G, Berrut G. [Frailty in older population: a brief position paper from the French society of geriatrics and gerontology]. Geriatr Psychol Neuropsychiatr Vieil. 2011 Dec;9(4):387-90. doi: 10.1684/pnv.2011.0311. French. PMID 22182814
- [Result] Has, " Comment repérer la fragilité en soins ambulatoires ? ", Points clés Solut. Organ. des Parcour., 2013.
- [Result] Studenski S, Perera S, Patel K, Rosano C, Faulkner K, Inzitari M, Brach J, Chandler J, Cawthon P, Connor EB, Nevitt M, Visser M, Kritchevsky S, Badinelli S, Harris T, Newman AB, Cauley J, Ferrucci L, Guralnik J. Gait speed and survival in older adults. JAMA. 2011 Jan 5;305(1):50-8. doi: 10.1001/jama.2010.1923. PMID 21205966
- [Result] Abellan van Kan G, Rolland Y, Andrieu S, Bauer J, Beauchet O, Bonnefoy M, Cesari M, Donini LM, Gillette Guyonnet S, Inzitari M, Nourhashemi F, Onder G, Ritz P, Salva A, Visser M, Vellas B. Gait speed at usual pace as a predictor of adverse outcomes in community-dwelling older people an International Academy on Nutrition and Aging (IANA) Task Force. J Nutr Health Aging. 2009 Dec;13(10):881-9. doi: 10.1007/s12603-009-0246-z. PMID 19924348
- [Result] Collard RM, Boter H, Schoevers RA, Oude Voshaar RC. Prevalence of frailty in community-dwelling older persons: a systematic review. J Am Geriatr Soc. 2012 Aug;60(8):1487-92. doi: 10.1111/j.1532-5415.2012.04054.x. Epub 2012 Aug 6. PMID 22881367
- [Result] A. Cherubini, L. Demougeot, A. Cruz Jentoft, A. Curgunlu, J. P. Michel, H. Roberts, A. Aihie Sayer, T. Strandberg, E. Topinkova, F. M. Trotta, D. Z. B. Van Asselt, B. Vellas, D. Zekry, et M. Cesari, " Relationship between the Gérontopole Frailty Screening Tool and the frailty phenotype in primary care ", Eur. Geriatr. Med., vol. 6, no 6, p. 518-522, 2015.
- [Result] Chiu AY, Au-Yeung SS, Lo SK. A comparison of four functional tests in discriminating fallers from non-fallers in older people. Disabil Rehabil. 2003 Jan 7;25(1):45-50. PMID 12554391
- [Result] Wrisley DM, Kumar NA. Functional gait assessment: concurrent, discriminative, and predictive validity in community-dwelling older adults. Phys Ther. 2010 May;90(5):761-73. doi: 10.2522/ptj.20090069. Epub 2010 Apr 1. PMID 20360052
- [Result] Smith, " Validation and Reliability of the Elderly Mobility Scale ", Physiotherapy, vol. 80 (11), no June 2012, p. 744-747, 1994.
- [Result] Thomas JI, Lane JV. A pilot study to explore the predictive validity of 4 measures of falls risk in frail elderly patients. Arch Phys Med Rehabil. 2005 Aug;86(8):1636-40. doi: 10.1016/j.apmr.2005.03.004. PMID 16084819